CLINICAL TRIAL: NCT07260734
Title: AUGMENTED RESPONSE OF VOLATILE BIOMARKERS IN THE ASSESSMENT OF OESOPHAGOGASTRIC CANCER (AROMA2)
Acronym: AROMA2
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 353374
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: OESOPHAGO-GASTRIC CARCINOMA; Oesophageal Adenocarcinoma; Gastric Adenocarcinoma and Gastroesophageal Junction Adenocarcinoma; Oesophageal Cancer Nos; Oesophageal Cancer; Oesophageal Junction Cancer; Breath Tests; Volatile Organic Compound
Keywords: Oesophageal adenocarcinoma; Gastric adenocarcinoma; Breath testing; Microbiome; Augmentation; Volatile Organic Compounds; Volatilomics; Breathomics
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Breath
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants referred along upper gastrointestinal suspected cancer pathways: Participants referred by GPs to secondary care for the reference test (i.e. upper gastrointestinal endoscopy, CT/MRI/ultrasound ± histological/cytology). Participants will be followed up (within 3 months) to determine whether they had a diagnosis of upper gastrointestinal adenocaricinoma or a normal/benign diagnosis.
  Interventions: Diagnostic Test: Breath Test

INTERVENTIONS:
Diagnostic Test: Breath Test — Diagnostic Test: Breath test Participants must be fasted for a minimum of six hours prior to breath sample collection. Breath samples will be collected prior to the reference test for each participant.
  Participants will then be asked to consume an Oral Stimulant Drink (OSD). The oral stimulant drink (120ml) will be composed of 25g glucose, 25g glycerol, 0.6g iron sulphate, 1.2g of "Thicken Up" thickener and combined amino acids (0.08g tyrosine, 1.8g phenylalanine, 2.1g glutamic acid).
  Diagnostic Test: Augmented breath test:
  Participants will then be asked to repeat a breath sample 15 minutes after consumption of the OSD.

SUMMARY:
Cancer of the stomach and oesophagus is among the world's top five cancers. Survival rates are very poor as the disease presents late and early symptoms are non-specific. The study team has developed a non-invasive test for cancers of the stomach and oesophagus based on the detection of volatile organic compounds in exhaled breath. These compounds are known to be produced by both cancers as well as cancer associated bacteria within the gut.

The proposed innovation is to improve the accuracy of this test by investigating whether simple metabolic substrates can increase the production of these volatile organic compounds by both the tumour and its associated bacteria.

DETAILED DESCRIPTION:
Oesophagogastric Cancer Early Detection: A Clinical Challenge

The detection of oesophagogastric cancer at an early stage remains an unmet clinical need. It's incidence in the UK and many other western countries has risen dramatically in recent years. Challenges in diagnosis are attributable to the largely non-specific nature of its early symptoms, which overlap with benign gastrointestinal conditions, alongside the resource intense and invasive nature of the current diagnostic pathways such as endoscopy. The so called 'red flag' symptoms that prompt more urgent investigation are often associated with advanced disease where curative treatments are limited. As a result, the five-year survival rate for oesophagogastric cancer in the UK remains distressingly low at 15-20%, one of the poorest in Europe. Early detection offers the best chance for effective intervention, where minimally invasive treatments and surgical procedures can lead to survival rates of over 85%.

There is a growing body of evidence that volatile organic compounds (VOCs), which are small molecules exhaled in breath, hold promise as non-invasive biomarkers for cancer detection in the form of a breath test. Our work suggests that VOCs are produced by both cancer cells and the tumour-associated microbiome. Our understanding of the pathways leading to VOC production allow us to propose augmentation of the breath test using certain nutrients to increase the production of volatile markers and improve the tests accuracy.

We have developed a breath test for diagnosing oesophagogastric cancer, starting with volatile biomarker discovery and progressing to a multi-centre NIHR-funded clinical study which demonstrated a sensitivity of 80% and specificity of 81%. To explore the origin of VOCs in oesophagogastric cancer, we developed an in-vivo human model that allowed for the compartmental measurement of VOCs from the gastrointestinal tract, airways, and mixed breath during general anaesthesia. The comparable levels of volatile fatty acids in both mixed and bronchial breath from cancer patients suggest that the primary source of these VOCs is the lungs, likely entering the breath through the systemic circulation.

Alongside this we have developed standardised operating procedures for VOC analysis with a platform for high-throughput breath analysis adherent to ISO accreditation standards. Our validated methodology has a VOC quantitation limit of 1.25 ng/L with established quality assurance and control procedures.

The AROMA programme is a comprehensive initiative aimed at understanding the pathways underpinning cancer-derived VOC production. Instead of only focusing on improving the sensitivity of detection equipment, our proposed solution involves augmenting the production of VOCs by introducing simple nutrients. These nutrients are anticipated to be metabolised rapidly by cancer cells and the cancer-associated microbiome to augment cancer-specific VOC production. By exploiting these VOC-pathways we will develop a breath test for oesophagogastric cancer that has a clinically acceptable sensitivity and specificity. After conducting optimisation experiments in a proof of principal study (AMNED; REC Ref:18/LO/0078), we developed an oral stimulant drink (OSD) composed of glucose, glycerol, amino acids and iron. The breath of patients with oesophagogastric cancer(n=30) and controls (n=30) was collected for 2 hours at 30-minute intervals after consuming the OSD. The peak VOC response varied but occurred within an hour of consumption. We also showed that VOC production by oesophagogastric cancer-associated bacteria could be enhanced using the same nutrient substrates.

In the AROMA1 study (n=648), a cancer detection model based on a breath test, augmented by an OSD, was developed. The AROMA Bioresource (n=335) established a comprehensive bioresource of tissue from cancer and non-cancer patients to understand pathways leading to VOC origin.

Justification for AROMA2

The AROMA2 study is a pivotal next step in this programme. AROMA2 will test the breath test in a multi-centre triple-blinded clinical trial, evaluating its sensitivity and specificity in patients referred to the upper gastrointestinal (GI) cancer pathway. These patients present with symptoms suggestive of upper GI cancer but have an unknown diagnosis. It will provide essential validation of the breath test in a real-world clinical setting, to establish the test's diagnostic accuracy in a clinical context.

Methods

At least 5400 individuals with suspected upper GI cancer, referred from primary care along upper gastrointestinal cancer pathways, will be recruited from 20+ centres. The aim is to have 216 cancers and 5184 controls with complete dataset (reliable breath data and results of reference test). Breath samples, before and after an oral stimulant drink (OSD), will be collected on thermal desorption tubes which will be analysed using gas chromatography-mass spectrometry (GC-MS). The diagnostic accuracy of breath test to detect cancer will be tested.

Anticipated impact and dissemination: The non-invasive breath test will provide direct patient benefit through earlier and accurate detection of Upper GI cancers, along with higher patient acceptability. Ensuring timely referral will translate to curative treatment and improved long-term survival. Outcomes will be disseminated via conference presentations, publications, the local public advisory group (PAG), charities, the local research website and social media.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old.
* Participants referred from primary care according to the urgent suspected cancer referral guidelines for potential underlying oesophagogastric cancer a for the reference test (described below).
* Willing and able to provide informed written consent to take part in study.

Exclusion Criteria:

* Previous oesophageal or gastric resection
* History of cancer within three years (other than non-melanoma skin cancers)
* Co-morbidities preventing breath collection
* Pregnant participants
* Allergies to any of the constituents of the nutrient drink including glucose, glycerol, iron sulphate, Maltodextrin (Corn, Potato), Xanthan Gum, Potassium Chloride, tyrosine, phenylalanine, and glutamic acid
* Unable or unwilling to provide informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18 years or over with suspected cancer, referred from primary care for further specialized investigations.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Validation of VOC biomakrer model for Upper GI Adenocarcinoma | 3 years
  GC-MS will be used to confirm the presence of upper gastrointestinal cancer-associated VOCs in order to validate the detection model developed in AROMA1

CONTACTS AND LOCATIONS:
Overall Officials: George Hanna, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: No
Participants will be offered to have study data shared with them on completion of the study

REFERENCES:
- See also: Related Info — https://www.thehannagroup.org/aroma/